CLINICAL TRIAL: NCT03435965
Title: Dilemma for Diagnosis of Amniotic Fluid Leakeage by AmnioQuickDuo+
Brief Title: PROM by AmnioQuick Duo+ in Egyptian Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aljazeera Hospital (Other)
Collaborators: Kasr El Aini Hospital (Other); National Research Centre, Egypt (Other)
Responsible Party: Principal Investigator, Mahmoud Alalfy, Assistant Researcher , National Research centre and Specialist of Obstetrics and Gynecology in Aljazeerah hospital, Aljazeera Hospital
Other Study IDs: PROM by AmnioQuick Duo+
Record Dates: First submitted 2018-02-10; First posted 2018-02-19 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: PROM (Pregnancy)
MeSH Terms: conditions — Fetal Membranes, Premature Rupture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PPROM from 20- less than 28 weeks: pregnant ladies with PROM from 20 - 28 weeks
  Interventions: Diagnostic Test: AmnioQuickDuo+
- PROM from more than 28 weeks - less than 37 weeks: pregnant ladies with PROM from more than 28- less than37 weeks
  Interventions: Diagnostic Test: AmnioQuickDuo+
- control group pregnant ladies in labour after 37 weeks: control group pregnant ladies in labour after 37 weeks with rupture of membrane in labour or in cs
  Interventions: Diagnostic Test: AmnioQuickDuo+

INTERVENTIONS:
Diagnostic Test: AmnioQuickDuo+ — AmnioQuickDuo+ kit for detection of PROM

SUMMARY:
Preterm premature rupture of the membranes (PPROM) is responsible for one-third of all preterm births. Optimum treatment relies on accurate diagnosis and gestational age. The diagnosis of PPROM is made by a combination of examination, patient history and some simple tests.

DETAILED DESCRIPTION:
Premature rupture of the fetal membranes (PROM) is the rupture of the amniotic membranes with release of the amniotic fluid prior to the onset of labour. PROM may be subdivided into term -PROM (TPROM, i.e. PROM after 37 weeks of gestation) and preterm PROM (PPROM, i.e. PROM prior to 37 weeks of gestation). PPROM occurs in approximately 3% of pregnancies and is responsible for a third of all preterm births.The diagnosis of PPROM is made by examination , patient history and simple testing. Patient history has an accuracy of 90% for the diagnosis of PPROM

ELIGIBILITY:
Inclusion Criteria:

* pregnant ladies with PROM from 20- 37 weeks

Exclusion Criteria:

* Gestational Age >37 wks Non reassuring CTG Signs of chorioamnonitis ( Fever , maternal or fetal tachycardia , Foul cervical discharge , uterine tenderness or high TLC ) Antepartum hemorrhage

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant ladies with PROM
Study Population: - pregnant ladies with PROM from 20- 37 weeks came to the hospital to confirm PROM
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-10-15 (Estimated); Study Completion 2019-11-01 (Estimated)

PRIMARY OUTCOMES:
number of participants who was diagnosed with leakage of liqour by AmnioQuickDuo+ | within a week
  the accuracy of amnioQuick to diagnose PROM

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Principal Investigator — Algazeerah hospital -Location (Giza -Egypt ) and National Research centre egypt
Locations (2):
- Egypt (2):
  - Kasralainy Hospital, Cairo
  - Algazeerah, Giza

IPD SHARING:
Plan to Share IPD: No
the data will be shared after finishing the research